CLINICAL TRIAL: NCT05451550
Title: Comparison of Effects and Safety in Providing Controlled Hypotension During Arthroscopic Shoulder Surgery Between General Anesthesia and General Anesthesia Combined With Nerve Block
Brief Title: The Effects of General Anesthesia and Combined Anesthesia in Controlled Hypotension During Arthroscopic Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gang202207
Record Dates: First submitted 2022-06-20; First posted 2022-07-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Shoulder Injuries; Shoulder Osteoarthritis
MeSH Terms: conditions — Shoulder Injuries | interventions — Brachial Plexus Block; Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia group (Experimental): Patients were maintained with propofol/remifentanil in general anesthesia
  Interventions: Procedure: General anesthesia
- General anesthesia combined with brachial plexus block group (Experimental): An additional ultrasound-guided brachial plexus block were performed
  Interventions: Procedure: Brachial plexus block; Procedure: General anesthesia
- general anesthesia combined with suprascapular nerve block group (Experimental): An additional ultrasound-guided suprascapular nerve block were performed
  Interventions: Procedure: General anesthesia; Procedure: Suprascapular nerve block

INTERVENTIONS:
Procedure: Brachial plexus block — An additional ultrasound-guided suprascapular nerve block(0.375% ropivacaine) were performed before general anesthesia induction in general anesthesia combined with brachial plexus block group
  Other Names: General anesthesia combined with brachial plexus block group
  Arms: General anesthesia combined with brachial plexus block group
Procedure: General anesthesia — General anesthesia were performed according to clinical routine: induction drugs: propofol, sufentanil, rocuronium, maintenance drugs: propofol, sevoflurane and remifentanil, Laryngeal mask ventilation.
Procedure: Suprascapular nerve block — An additional ultrasound-guided suprascapular nerve block(0.375% ropivacaine) were performed before general anesthesia induction in general anesthesia combined with brachial plexus block group
  Other Names: General anesthesia combined with suprascapular nerve block group
  Arms: general anesthesia combined with suprascapular nerve block group

SUMMARY:
Controlled hypotension is one of the important techniques used for facilitates the clarity of the surgical field during arthroscopic shoulder surgery. Brachial plexus or its branches block provides excellent analgesia during arthroscopic shoulder surgery. To test the hypothesis that, during arthroscopic shoulder surgery, general anesthesia combined with nerve block could provide more stable hemodynamic index than general anesthesia. Patients undergoing arthroscopic shoulder surgery were enrolled and divided into 3 groups: general anesthesia group, general anesthesia combined with brachial plexus block, and general anesthesia combined with suprascapular nerve block group. The dosage of vasoactive drugs and anesthetics, parameters of perioperative bleeding, hemodynamic parameters, systemic oxygen metabolism, kidney functions, as well as procedure process and postoperative adverse reactions were recorded and compared between the groups.

DETAILED DESCRIPTION:
Controlled hypotension is one of the important techniques used for minimizing bleeding and facilitates the clarity of the surgical field during arthroscopic shoulder surgery. Although surgical field visualization is important in arthroscopic shoulder surgery, the complications associated with controlled hypotension for surgery should be considered. The implementation of controlled hypotension requires a large amount of antihypertensive agents or anesthetics, it may cause instability of the circulatory system, organ hypoperfusion, or subsequent ischemic injury. Brachial plexus or its branches block provides excellent analgesia during arthroscopic shoulder surgery. However, few data are currently available in the literature evaluating brachial plexus or its branches block and controlled hypotension during arthroscopic shoulder surgery. To obtain more information on this topic, the investigators conducted this prospective randomized study to test the hypothesis that, during arthroscopic shoulder surgery, general anesthesia combined with nerve block could provide more stable hemodynamic index than general anesthesia.

Methods:

The inclusion criteria are (1) planned elective arthroscopic shoulder surgery, need controlled hypotension under general anesthesia; (2) aged 60-75 years; (3) ASA grade II or III; and (4) estimated operative time < 120 min. The exclusion criteria were (1) preoperative blood pressure systolic ≥ 160 mmHg or diastolic ≥ 100 mmHg or pulse pressure ≥ 60 mmHg; (2) comorbidities of severe cardiovascular disease, including cardiac function grade III or IV, severe aortic stenosis, aortic valve insufficiency, severe coronary heart disease, bradycardia, and atrioventricular block above degree I; (3) history of cerebral infarction, Alzheimer's disease, or cerebrovascular incident; (4) liver and/or kidney dysfunction; (5) severe anemia, shock, hypovolemia, or respiratory dysfunction; (6) previous history of phlebitis or thrombosis, closed-angle glaucoma; and (7) BMI > 25 or < 18. Patients with intraoperative blood loss > 1500 mL or operation time > 4 h would be further excluded from the analysis.

The included patients were divided into 3 groups: general anesthesia group, general anesthesia combined with brachial plexus block, and general anesthesia combined with suprascapular nerve block group. For controlled hypotension during surgery, all patients were maintained with propofol/remifentanil in general anesthesia. An additional ultrasound-guided brachial plexus block or suprascapular nerve block were performed in general anesthesia combined with brachial plexus block or general anesthesia combined with suprascapular nerve block group. The dose of each agent was adjusted to maintain the mean arterial blood pressure (MAP) at 60 to 70 mm Hg and the BIS at 40 to 60. nicardipine and phenylephrine served mainly to control the target MAP, Norepinephrine and esmolol were also used as needed.

The dosage of vasoactive drugs (vasopressor-inotrope dose was calculated by adding norepinephrine equivalents of total norepinephrine, epinephrine, phenylephrine, and vasopressin dose used during surgery, using the following formula: total vasopressor-inotrope dose = [norepinephrine (µg/min) × min] + [epinephrine (µg/min) × min] + [(phenylephrine (µg/min) ×min) ÷ 10] + [vasopressin (U/h) × 8.33 × min]) and anesthetics, parameters of perioperative bleeding, hemodynamic parameters(blood pressure, heart rate, pulse oximetry), systemic oxygen metabolism, kidney functions, as well as procedure process and postoperative adverse reactions were recorded and compared between the groups. The incidence of postoperative complications (within 7 days, such as Organ dysfunction) were also recorded.

Statistical analysis and get conclusions.

ELIGIBILITY:
Inclusion Criteria:

* (1) planned elective arthroscopic shoulder surgery, need controlled hypotension under general anesthesia; (2) aged 60-75 years; (3) ASA grade II or III; and (4) estimated operative time < 120 min.

Exclusion Criteria:

* (1) preoperative blood pressure systolic ≥ 160 mmHg or diastolic ≥ 100 mmHg or pulse pressure ≥ 60 mmHg; (2) comorbidities of severe cardiovascular disease, including cardiac function grade III or IV, severe aortic stenosis, aortic valve insufficiency, severe coronary heart disease, bradycardia, and atrioventricular block above degree I; (3) history of cerebral infarction, Alzheimer's disease, or cerebrovascular incident; (4) liver and/or kidney dysfunction; (5) severe anemia, shock, hypovolemia, or respiratory dysfunction; (6) previous history of phlebitis or thrombosis, closed-angle glaucoma; and (7) BMI > 25 or < 18. Patients with intraoperative blood loss > 1500 mL or operation time > 4 h would be further excluded from the analysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-17 (Estimated); Primary Completion 2024-09-29 (Estimated); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
The dosage of total vasopressor-inotrope dose between groups | 1 day
  The dosage of total vasopressor-inotrope dose (Calculate by formula) between the groups

SECONDARY OUTCOMES:
The dosage of anesthetics between groups | 1 day
  The dosage of propofol(milligram) and sevoflurane(milliliter) between groups
Blood pressure between the groups | 1 day
  Blood pressure(millimeter of mercury) between the groups
The incidence of postoperative complications | 3 day
  The incidence of postoperative complications (within 7 days, such as Organ dysfunction) between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No